CLINICAL TRIAL: NCT03939598
Title: Feasibility of Preoperative Tattooing of Percutaneously Biopsied Axillary Lymph Node: A Quasi Experimental Pilot Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Abida K. Sattar, MD, FACS, Chief of Breast Surgery, Aga Khan University
Other Study IDs: 2018-0345-1105
Record Dates: First submitted 2019-04-24; First posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Breast Neoplasm
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates utility of a novel technique using India Ink to aid in the identification and retrieval of axillary lymph nodes during surgery, in breast cancer patients with suspicious lymph nodes.

The first part of the study will evaluate the feasibility of the technique in patients who commence their treatment with surgery. Provided its success, the second part of the study will evaluate the applicability of this same technique in patients who receive chemotherapy before having surgery.

DETAILED DESCRIPTION:
Breast cancer is the leading cause of cancer mortality among females. Sentinel lymph node biopsy helps avoid axillary lymph node dissection and the associated morbidity. However, its utility is unclear in patients with biopsy proven axillary disease that has been treated with neoadjuvant chemotherapy. The objective of our study is to evaluate a) the feasibility of a novel technique of preoperatively tattooing suspicious lymph nodes with India ink, their intraoperative identification and retrieval in patients undergoing upfront breast and axillary surgery(Phase I); and b) the application of this technique in patients who undergo surgery after receiving neo-adjuvant chemotherapy i.e. lag time between tattooing and lymph node retrieval (Phase II) with the ultimate objective to see if the status of the excised sentinel and tattooed lymph node will be predictive of the status of the axilla.

A quasi-experimental pilot study will be conducted to evaluate the feasibility of tattooing suspicious lymph nodes with sterile black India ink. The study will be conducted in two phases, with the second phase conditional upon the successful results of the first. In Phase I, only 10 patients who are committed to undergo upfront surgery (without neoadjuvant chemotherapy) will be included. These patients will have the suspicious lymph node tattooed by injecting India ink at the time of ultrasound guided core needle biopsy. Intraoperatively, the axilla will be inspected to determine whether India ink tattooed in the lymph nodes can be visualized by the surgeon. Microscopic inspection for the presence of the dye in nodes retrieved by sentinel biopsy and/or axillary dissection will also be done. In Phase II, this process will be repeated for patients who undergo surgery after neoadjuvant chemotherapy and concordance between the sentinel, tattooed and non-sentinel nodes will be determined.

Ethical approval was obtained from the Aga Khan University Ethical Review Board (ERC# 2018-0345-1105). The process of sentinel node biopsy is a safe and routinely performed procedure at our institution. Intradermal injection of methylene blue can lead to skin necrosis; intra-parenchymal injection can cause induration and erythema with associated pain. These side effects can be minimized by diluting methylene blue which will be done. The complications that can result from all additional steps of study procedures will be discussed with the patient and their full responsibility will be borne by the institution. Although sterile black India Ink is safe to administer but possible side effects can include mucosal inflammation due to spillage of the ink, abscess formation and others such as an allergic reaction. If any of these situations are encountered full responsibility to treat the side effects will be borne by the study team using departmental funds.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patient (biopsy proven or clinically suspected) with clinically suspicious (palpable on clinical exam or abnormal by ultrasound criteria but not biopsied yet) ipsilateral axillary lymph node(s). The ultrasonographic examination will be considered suspicious for metastasis if one or more of following criteria are present: 1. Eccentric cortical enlargement (>3 mm) or lobulation with displacement of hilum 2. Absent hilum and irregular border and hypoechoic echotexture 3. Spherical node 4. Perinodal vascularity. (18-20)
* Participants willing to undergo axillary lymph node percutaneous biopsy with marking/tattooing of the biopsied lymph node at AKUH
* Participants intending to have definitive surgery at AKUH

Exclusion Criteria:

* Participants with terminal disease like renal failure will be excluded because these conditions can have profound effect on their course of treatment
* Participants with distant metastases
* Participants with prior breast or axillary surgery
* Participants with bilateral breast cancer, and those who have already had an axillary core needle biopsy prior to inclusion (to avoid a second procedure for tattooing)
* Participants with recurrent breast malignancy because their course of treatment might be different
* Participants that were initially suspected to have breast cancer, but pathology results did not confirm the diagnosis
* Pregnant and lactating women
* Men with breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients reporting to Breast Surgery Clinic at Aga Khan University, Main Campus in Karachi, Pakistan
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-03-27 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Intra-operative identification of tattooed lymph node(s) in upfront surgery group (Phase I) | December 31, 2019
  In patients undergoing upfront surgery: The rate of successful intraoperative identification of axillary lymph nodes tattooed with black India ink preoperatively.
Intra-operative identification of tattooed lymph node(s) in the post-neoadjuvant surgery group (Phase II) | December 31, 2020
  In patients undergoing surgery post-neoadjuvant chemotherapy (and associated lag time): The rate of successful intraoperative identification of axillary lymph nodes tattooed with black India ink preoperatively.

SECONDARY OUTCOMES:
Concordance rate between identified sentinel node(s) and tattooed lymph node(s) | December 31, 2020
  The rate of concordance between the intra-operatively identified sentinel node and tattooed node(s)

CONTACTS AND LOCATIONS:
Overall Officials: Abida K. Sattar, MD, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Caudle AS, Cupp JA, Kuerer HM. Management of axillary disease. Surg Oncol Clin N Am. 2014 Jul;23(3):473-86. doi: 10.1016/j.soc.2014.03.007. Epub 2014 Apr 13. PMID 24882346
- [Background] Krag DN, Anderson SJ, Julian TB, Brown AM, Harlow SP, Ashikaga T, Weaver DL, Miller BJ, Jalovec LM, Frazier TG, Noyes RD, Robidoux A, Scarth HM, Mammolito DM, McCready DR, Mamounas EP, Costantino JP, Wolmark N; National Surgical Adjuvant Breast and Bowel Project. Technical outcomes of sentinel-lymph-node resection and conventional axillary-lymph-node dissection in patients with clinically node-negative breast cancer: results from the NSABP B-32 randomised phase III trial. Lancet Oncol. 2007 Oct;8(10):881-8. doi: 10.1016/S1470-2045(07)70278-4. PMID 17851130
- [Background] Krag DN, Anderson SJ, Julian TB, Brown AM, Harlow SP, Costantino JP, Ashikaga T, Weaver DL, Mamounas EP, Jalovec LM, Frazier TG, Noyes RD, Robidoux A, Scarth HM, Wolmark N. Sentinel-lymph-node resection compared with conventional axillary-lymph-node dissection in clinically node-negative patients with breast cancer: overall survival findings from the NSABP B-32 randomised phase 3 trial. Lancet Oncol. 2010 Oct;11(10):927-33. doi: 10.1016/S1470-2045(10)70207-2. PMID 20863759
- [Background] Fisher B, Jeong JH, Anderson S, Bryant J, Fisher ER, Wolmark N. Twenty-five-year follow-up of a randomized trial comparing radical mastectomy, total mastectomy, and total mastectomy followed by irradiation. N Engl J Med. 2002 Aug 22;347(8):567-75. doi: 10.1056/NEJMoa020128. PMID 12192016
- [Background] Giuliano AE, Ballman K, McCall L, Beitsch P, Whitworth PW, Blumencranz P, Leitch AM, Saha S, Morrow M, Hunt KK. Locoregional Recurrence After Sentinel Lymph Node Dissection With or Without Axillary Dissection in Patients With Sentinel Lymph Node Metastases: Long-term Follow-up From the American College of Surgeons Oncology Group (Alliance) ACOSOG Z0011 Randomized Trial. Ann Surg. 2016 Sep;264(3):413-20. doi: 10.1097/SLA.0000000000001863. PMID 27513155
- [Background] Pilewskie M, Morrow M. Axillary Nodal Management Following Neoadjuvant Chemotherapy: A Review. JAMA Oncol. 2017 Apr 1;3(4):549-555. doi: 10.1001/jamaoncol.2016.4163. PMID 27918753
- [Background] Caudle AS, Yang WT, Krishnamurthy S, Mittendorf EA, Black DM, Gilcrease MZ, Bedrosian I, Hobbs BP, DeSnyder SM, Hwang RF, Adrada BE, Shaitelman SF, Chavez-MacGregor M, Smith BD, Candelaria RP, Babiera GV, Dogan BE, Santiago L, Hunt KK, Kuerer HM. Improved Axillary Evaluation Following Neoadjuvant Therapy for Patients With Node-Positive Breast Cancer Using Selective Evaluation of Clipped Nodes: Implementation of Targeted Axillary Dissection. J Clin Oncol. 2016 Apr 1;34(10):1072-8. doi: 10.1200/JCO.2015.64.0094. Epub 2016 Jan 25. PMID 26811528
- [Background] Kuehn T, Bauerfeind I, Fehm T, Fleige B, Hausschild M, Helms G, Lebeau A, Liedtke C, von Minckwitz G, Nekljudova V, Schmatloch S, Schrenk P, Staebler A, Untch M. Sentinel-lymph-node biopsy in patients with breast cancer before and after neoadjuvant chemotherapy (SENTINA): a prospective, multicentre cohort study. Lancet Oncol. 2013 Jun;14(7):609-18. doi: 10.1016/S1470-2045(13)70166-9. Epub 2013 May 15. PMID 23683750
- [Background] Boughey JC, Suman VJ, Mittendorf EA, Ahrendt GM, Wilke LG, Taback B, Leitch AM, Kuerer HM, Bowling M, Flippo-Morton TS, Byrd DR, Ollila DW, Julian TB, McLaughlin SA, McCall L, Symmans WF, Le-Petross HT, Haffty BG, Buchholz TA, Nelson H, Hunt KK; Alliance for Clinical Trials in Oncology. Sentinel lymph node surgery after neoadjuvant chemotherapy in patients with node-positive breast cancer: the ACOSOG Z1071 (Alliance) clinical trial. JAMA. 2013 Oct 9;310(14):1455-61. doi: 10.1001/jama.2013.278932. PMID 24101169
- [Background] Bryant JA, Siddiqi NJ, Loveday EJ, Irvine GH. Presurgical, ultrasound-guided anchor-wire marking of impalpable cervical lymph nodes. J Laryngol Otol. 2005 Aug;119(8):627-8. doi: 10.1258/0022215054516241. PMID 16102218
- [Background] Straver ME, Loo CE, Alderliesten T, Rutgers EJ, Vrancken Peeters MT. Marking the axilla with radioactive iodine seeds (MARI procedure) may reduce the need for axillary dissection after neoadjuvant chemotherapy for breast cancer. Br J Surg. 2010 Aug;97(8):1226-31. doi: 10.1002/bjs.7073. PMID 20602508
- [Background] Donker M, Straver ME, Wesseling J, Loo CE, Schot M, Drukker CA, van Tinteren H, Sonke GS, Rutgers EJ, Vrancken Peeters MJ. Marking axillary lymph nodes with radioactive iodine seeds for axillary staging after neoadjuvant systemic treatment in breast cancer patients: the MARI procedure. Ann Surg. 2015 Feb;261(2):378-82. doi: 10.1097/SLA.0000000000000558. PMID 24743607
- [Background] Choy N, Lipson J, Porter C, Ozawa M, Kieryn A, Pal S, Kao J, Trinh L, Wheeler A, Ikeda D, Jensen K, Allison K, Wapnir I. Initial results with preoperative tattooing of biopsied axillary lymph nodes and correlation to sentinel lymph nodes in breast cancer patients. Ann Surg Oncol. 2015 Feb;22(2):377-82. doi: 10.1245/s10434-014-4034-6. Epub 2014 Aug 28. PMID 25164040
- [Background] Caudle AS, Yang WT, Mittendorf EA, Black DM, Hwang R, Hobbs B, Hunt KK, Krishnamurthy S, Kuerer HM. Selective surgical localization of axillary lymph nodes containing metastases in patients with breast cancer: a prospective feasibility trial. JAMA Surg. 2015 Feb;150(2):137-43. doi: 10.1001/jamasurg.2014.1086. PMID 25517573
- [Background] Park S, Koo JS, Kim GM, Sohn J, Kim SI, Cho YU, Park BW, Park VY, Yoon JH, Moon HJ, Kim MJ, Kim EK. Feasibility of Charcoal Tattooing of Cytology-Proven Metastatic Axillary Lymph Node at Diagnosis and Sentinel Lymph Node Biopsy after Neoadjuvant Chemotherapy in Breast Cancer Patients. Cancer Res Treat. 2018 Jul;50(3):801-812. doi: 10.4143/crt.2017.210. Epub 2017 Aug 17. PMID 28814071
- [Background] Trakarnsanga A, Akaraviputh T. Endoscopic tattooing of colorectal lesions: Is it a risk-free procedure? World J Gastrointest Endosc. 2011 Dec 16;3(12):256-60. doi: 10.4253/wjge.v3.i12.256. PMID 22195235
- [Background] Holwitt DM, Swatske ME, Gillanders WE, Monsees BS, Gao F, Aft RL, Eberlein TJ, Margenthaler JA. Scientific Presentation Award: The combination of axillary ultrasound and ultrasound-guided biopsy is an accurate predictor of axillary stage in clinically node-negative breast cancer patients. Am J Surg. 2008 Oct;196(4):477-82. doi: 10.1016/j.amjsurg.2008.06.006. Epub 2008 Aug 23. PMID 18723153
- [Background] Oz A, Demirkazik FB, Akpinar MG, Soygur I, Baykal A, Onder SC, Uner A. Efficiency of ultrasound and ultrasound-guided fine needle aspiration cytology in preoperative assessment of axillary lymph node metastases in breast cancer. J Breast Cancer. 2012 Jun;15(2):211-7. doi: 10.4048/jbc.2012.15.2.211. Epub 2012 Jun 28. PMID 22807939
- [Background] Deurloo EE, Tanis PJ, Gilhuijs KG, Muller SH, Kroger R, Peterse JL, Rutgers EJ, Valdes Olmos R, Schultze Kool LJ. Reduction in the number of sentinel lymph node procedures by preoperative ultrasonography of the axilla in breast cancer. Eur J Cancer. 2003 May;39(8):1068-73. doi: 10.1016/s0959-8049(02)00748-7. PMID 12736105
- [Derived] Sattar AK, Ali B, Masroor I, Afzal S, Tariq MU, Idrees R, Uzzaman M, Khalid W. Feasibility of preoperative tattooing of percutaneously biopsied axillary lymph node: an experimental pilot study. Pilot Feasibility Stud. 2020 Sep 24;6:140. doi: 10.1186/s40814-020-00682-2. eCollection 2020. PMID 32983557

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-27): https://cdn.clinicaltrials.gov/large-docs/98/NCT03939598/Prot_SAP_000.pdf